CLINICAL TRIAL: NCT07383740
Title: Test-Retest Reliability of a Submaximal Exercise Test in Patients With Hip- and/or Knee Osteoarthritis
Brief Title: Test-Retest Reliability of a Submaximal Exercise Test in Patients With Hip and Knee Osteoarthritis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Test-retest_adapted_EB
Record Dates: First submitted 2026-01-19; First posted 2026-02-03 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Osteo Arthritis Knee and Hip
Keywords: Osteoarthritis; knee osteoarthritis; hip osteoarthritis; exercise test; reliability; cardiorespiratory fitness; test-retest
MeSH Terms: conditions — Osteoarthritis; Osteoarthritis, Knee; Osteoarthritis, Hip

STUDY DESIGN:
Intervention Model Description: Test-retest reliability of a submaximal cycle ergometer test.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Forty patients with osteoarthritis in hip or knee (Experimental): Forty patients with hip or knee osteoarthritis on the waiting list for usual rehabilitation care will be recruited. The patientes will be screened for contraindications, and, if eligible, will complete a submaximal cycle ergometer test twice within one week.
  Interventions: Procedure: Submaximal cycle ergometer test-retest

INTERVENTIONS:
Procedure: Submaximal cycle ergometer test-retest — Performing a submaximal cycle ergometer test twice

SUMMARY:
The aim is to evaluate the test-retest reliability of the primary care-adapted Ekblom-Bak submaximal ergometer bicycle test in patients with hip- and/or knee osteoarthritis (OA).

Forty patients with hip- and/or knee OA eligible for the Swedish national OA treatment program in primary care are to be recruited. After screening for contraindications, participants will perform the aEB-test twice within 1-2 weeks.

The investigators hypothezise that the test will demonstrate acceptable test-retest reliability in patients with hip- and/or knee OA.

To establish reliability is essential for future studies using this test in this population and may support its integration into routine clinical assessment.

ELIGIBILITY:
Inclusion Criteria:

* Currently listed on the waiting list for an osteoarthritis rehabilitation program due to clinically diagnosed hip and/or knee osteoarthritis.

Exclusion Criteria:

* Another primary cause of symptoms or disability, such as inflammatory joint disease or fracture.
* Another condition currently causing more symptoms than osteoarthritis, for example fibromyalgia.
* Insufficient understanding of written and spoken Swedish.
* Medication that affects heart rate.
* Contraindications for a submaximal ergometer bicycle test according to the screening protocol, such as heart disease.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male or female
Enrollment: 40 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Estimated VO2-max value. | Time between first and second submaximal cycle ergometer test should be one week.
  An estimated VO2-max value is obtained by performing the Ekblom Bak submaximal cycle ergometer test.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.researchweb.org/is/vgr/project/285943